CLINICAL TRIAL: NCT02600351
Title: A Phase 3b, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Ledipasvir/Sofosbuvir, With or Without Ribavirin, in HCV Infected Subjects Who Have Failed Prior Treatment With Sofosbuvir-based Therapies
Brief Title: Efficacy and Safety of Ledipasvir/Sofosbuvir, With or Without Ribavirin, in HCV Infected Participants Who Have Failed Prior Treatment With Sofosbuvir-based Therapies
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to lack of feasibility of enrolling participants, the study was terminated early.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1746
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Results first posted 2018-04-11 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C Virus (HCV); Ledipasvir/Sofosbuvir; Ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- LDV/SOF 12 weeks, without cirrhosis (Experimental): LDV/SOF for 12 weeks
  Interventions: Drug: LDV/SOF
- LDV/SOF + RBV 12 weeks, without cirrhosis (Experimental): LDV/SOF + RBV for 12 weeks
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF + RBV 12 weeks, with compensated cirrhosis (Experimental): LDV/SOF + RBV for 12 weeks
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 24 weeks, with compensated cirrhosis (Experimental): LDV/SOF for 24 weeks
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — Tablets administered orally in a divided daily dose according to weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF + RBV 12 weeks, with compensated cirrhosis; LDV/SOF + RBV 12 weeks, without cirrhosis

SUMMARY:
The primary objective of this study is to evaluate the efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed dose combination (FDC) for 12 weeks with or without ribavirin (RBV) in participants without cirrhosis, and LDV/SOF FDC for 12 weeks with RBV or LDV/SOF FDC for 24 weeks without RBV in participants with cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

* HCV RNA > 15 IU/mL at screening
* HCV genotype 1 or 4
* Chronic HCV infection (≥ 6 months)
* Prior virologic failure after treatment with SOF in combination with simeprevir (SMV) ± RBV or with RBV ± pegylated interferon (PEG)
* Cirrhotic and non-cirrhotic as determined by standard methods
* Male and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception

Key Exclusion Criteria:

* Prior exposure to approved or experimental non-structural protein (NS5A) inhibitors
* Prior exposure to nucleos(t)ide polymerase inhibitors, other than SOF
* Pregnant or nursing female or male with pregnant female partner
* Coinfection with HIV or hepatitis B virus
* Current or prior history of clinical hepatic decompensation
* Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with individual's treatment, assessment or compliance with the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (37):
- United States (34):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Pasadena, California
  - Rialto, California
  - Sacramento, California
  - Ventura, California
  - New Haven, Connecticut
  - Largo, Florida
  - Weston, Florida
  - Chicago, Illinois
  - Skokie, Illinois
  - Baltimore, Maryland
  - Columbia, Maryland
  - Worcester, Massachusetts
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Egg Harbor, New Jersey
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Seattle, Washington
- Canada (2):
  - Vancouver, British Columbia
  - Montreal, Quebec
- Ponce, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Tam E, Brown RS, Satapathy S, Shen X, Camus G, Copans A, et al. Efficacy and Safety of Ledipasvir/Sofosbuvir (LDV/SOF), with or without Ribavirin (RBV), for Treatment of HCV-mono and HIV/HCV Co-infected Patients Who Have Failed Prior Treatment with Non-NS5A, SOF-based Therapies [Poster THU-265]. The International Liver Congress™ 2017: European Association for the Study of the Liver (EASL); 2017 19-23 April; Amsterdam, the Netherlands.
- [Result] Tam E, Mantry PS, Satapathy SK, Ghali P, Shen X, Han LL, et al. A Phase 3b, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Ledipasvir/Sofosbuvir (LDV/SOF), with or without Ribavirin (RBV), in HCV Infected Subjects Who Have Failed Prior Treatment with Non-NS5A, SOF-based Therapies (RESCUE) [Poster PP0217]. Asian Pacific Association for the Study of the Liver (APASL); 2017 15-19 February; Shanghai, China.
- [Result] Tam E, Brown RS, Satapathy S, Camus G, Copans A, Rossaro L, et al. Ledipasvir/Sofosbuvir ± Ribavirin in HCV and HIV/HCV Prior SOF-based Virologic Failures (RESCUE and ACTG A5348 Studies) [Poster 568LB]. Conference on Retroviruses and Opportunistic Infections (CROI); 2017 13-16 February; Seattle, WA.
- [Result] Tam E, Luetkemeyer AF, Mantry PS, Satapathy SK, Ghali P, Kang M, Haubrich R, Shen X, Ni L, Camus G, Copans A, Rossaro L, Guyer B, Brown RS Jr; RESCUE and ACTG A5348 study investigators. Ledipasvir/sofosbuvir for treatment of hepatitis C virus in sofosbuvir-experienced, NS5A treatment-naive patients: Findings from two randomized trials. Liver Int. 2018 Jun;38(6):1010-1021. doi: 10.1111/liv.13616. Epub 2017 Dec 5. PMID 29091342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States (including a site in Puerto Rico), and Canada. The first participant was screened on 11 November 2015. The last study visit occurred on 29 May 2017.
Pre-assignment Details: 120 participants were screened.
Groups:
- LDV/SOF 12 Weeks, Without Cirrhosis: Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks in participants without cirrhosis
- LDV/SOF + RBV 12 Weeks, Without Cirrhosis: LDV/SOF (90/400 mg) FDC tablet orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks in participants without cirrhosis
- LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis: LDV/SOF (90 mg/400 mg) FDC tablet orally once daily + RBV (1000 or 1200 mg/day divided twice daily) for 12 weeks in participants with compensated cirrhosis
- LDV/SOF 24 Weeks, With Compensated Cirrhosis: LDV/SOF (90/400 mg) FDC tablet orally once daily for 24 weeks in participants with compensated cirrhosis
Period: Overall Study
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis
Started | 17 | 17 | 26 | 27
Completed | 12 | 17 | 20 | 22
Not Completed | 5 | 0 | 6 | 5
Not completed — Lack of Efficacy | 3 | 0 | 5 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Randomized but Not Treated | 1 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of study drug
Groups:
- LDV/SOF 12 Weeks, Without Cirrhosis: LDV/SOF (90/400 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks in participants without cirrhosis
- LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis: LDV/SOF FDC (90 mg/400 mg) tablet orally once daily + RBV (1000 or 1200 mg/day divided twice daily) for 12 weeks in participants with compensated cirrhosis
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis | Total
Number analyzed (Participants) | 16 | 17 | 25 | 24 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (5.7) | 57 (5.5) | 58 (7.8) | 60 (4.5) | 59 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 6 | 5 | 21
  Male | 10 | 13 | 19 | 19 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Black or African American | 6 | 5 | 6 | 3 | 20
  Other | 0 | 0 | 1 | 1 | 2
  White | 10 | 11 | 18 | 19 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 4 | 7 | 16
  Not Hispanic or Latino | 14 | 14 | 21 | 17 | 66
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 2 | 2 | 7 | 12
  Puerto Rico | 1 | 1 | 0 | 1 | 3
  United States | 14 | 14 | 23 | 16 | 67
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 1 | 2 | 0 | 1 | 4
    CT | 12 | 11 | 16 | 17 | 56
    TT | 3 | 4 | 9 | 6 | 22
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.45) | 6.4 (0.48) | 6.1 (0.59) | 6.0 (0.89) | 6.2 (0.67)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 1 | 4 | 7 | 8 | 20
  ≥ 800,000 IU/mL | 15 | 13 | 18 | 16 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Cessation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, < 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set by Actual Treatment: participants were grouped according to their cirrhotic status and the treatment/duration they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- LDV/SOF 12 Weeks, Without Cirrhosis: LDV/SOF (90/400 mg) FDC tablet orally once daily for 12 weeks in participants without cirrhosis
- LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis: LDV/SOF (90/400 mg) FDC tablet orally once daily + RBV (1000 or 1200 mg/day divided twice daily) for 12 weeks in participants with compensated cirrhosis
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis
Number analyzed (Participants) | 16 | 17 | 25 | 24
percentage of participants | 81.3 [54.4 to 96.0] | 100.0 [80.5 to 100.0] | 80.0 [59.3 to 93.2] | 91.7 [73.0 to 99.0]
Statistical Analysis 1: Comparison: LDV/SOF 12 Weeks, Without Cirrhosis vs LDV/SOF + RBV 12 Weeks, Without Cirrhosis; Test type: Non-Inferiority — With a 10% non-inferiority margin, a sample size of 90 participants per treatment group was required to provide at least 90% power to establish non-inferiority at the 1-sided 0.025 level, assuming the SVR12 rates were 98% for both groups; p = 0.065, Cochran-Mantel-Haenszel; Difference in percentages = -18.8, 95% CI 2-sided [-40.7 to 3.2]
Statistical Analysis 2: Comparison: LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis vs LDV/SOF 24 Weeks, With Compensated Cirrhosis; Test type: Non-Inferiority — With a 10% non-inferiority margin, a sample size of 125 participants per treatment group was required to provide at least 90% power to establish non-inferiority at the 1-sided 0.025 level, assuming the SVR12 rates were 95% for both groups; p = 0.25, Cochran-Mantel-Haenszel; Difference in percentages = -11.7, 95% CI 2-sided [-32.1 to 8.8]

2. Primary Outcome: Percentage of Participants Who Discontinued From Study Treatment for an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis
Number analyzed (Participants) | 16 | 17 | 25 | 24
percentage of participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With HCV RNA < the Lower Limit of Quantitation (LLOQ) at 4 and 24 Weeks Posttreatment
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set by Actual Treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis
Number analyzed (Participants) | 16 | 17 | 25 | 24
percentage of participants
  SVR4 | 93.8 [69.8 to 99.8] | 100.0 [80.5 to 100.0] | 88.0 [68.8 to 97.5] | 95.8 [78.9 to 99.9]
  SVR24 | 81.3 [54.4 to 96.0] | 100.0 [80.5 to 100.0] | 80.0 [59.3 to 93.2] | 91.7 [73.0 to 99.0]

4. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while receiving treatment.
Time Frame: Up to 24 weeks
Population: Full Analysis Set by Actual Treatment
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis
Number analyzed (Participants) | 16 | 17 | 25 | 24
percentage of participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA <LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set by Actual Treatment
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis
Number analyzed (Participants) | 16 | 17 | 25 | 24
percentage of participants | 18.8 | 0 | 20.0 | 8.3

6. Secondary Outcome: Number of Participants With Emerging Resistance
Description: The full-length NS3, NS5A, and NS5B coding regions were deep sequenced at pretreatment (baseline) for all participants included in the Full Analysis Set, and at posttreatment for all participants who relapsed.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set by Actual Treatment who have pre-existing NS5B, NS5A, and NS3/4A resistance-associated variants (RAVs) at baseline and who experienced virologic failure were analyzed. There were no participants with pre-existing RAVs who experienced virologic failure in the LDV/SOF+RBV 12 weeks, without cirrhosis group.
Measure: Count of Participants; unit: Participants
Groups:
- LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis: LDV/SOF FDC (90/400 mg) tablet orally once daily + RBV (1000 or 1200 mg/day divided twice daily) for 12 weeks in participants with compensated cirrhosis
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis
Number analyzed (Participants) | 3 | 0 | 5 | 2
Participants | 3 |  | 5 | 2

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | LDV/SOF 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, Without Cirrhosis | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis | LDV/SOF 24 Weeks, With Compensated Cirrhosis
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/25 | 1/24
Other Adverse Events (participants affected / at risk) | 11/16 | 14/17 | 19/25 | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks, Without Cirrhosis (N=16) | LDV/SOF + RBV 12 Weeks, Without Cirrhosis (N=17) | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis (N=25) | LDV/SOF 24 Weeks, With Compensated Cirrhosis (N=24)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks, Without Cirrhosis (N=16) | LDV/SOF + RBV 12 Weeks, Without Cirrhosis (N=17) | LDV/SOF + RBV 12 Weeks, With Compensated Cirrhosis (N=25) | LDV/SOF 24 Weeks, With Compensated Cirrhosis (N=24)
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Chills (General disorders) | 0 | 2 | 0 | 2
Fatigue (General disorders) | 2 | 6 | 7 | 4
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 5 | 2 | 9 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 5 | 3 | 3
Irritability (Psychiatric disorders) | 1 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 5 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to lack of feasibility of enrolling participants, the study was terminated early. Although, the non-inferiority tests were performed, the actual sample size was inadequate compared to the planned enrollment of 430 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2015-03-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT02600351/Prot_004.pdf
  • Study Protocol: Amendment 1 (2015-06-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02600351/Prot_005.pdf
  • Study Protocol: Amendment 2 (2015-07-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02600351/Prot_006.pdf
  • Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT02600351/SAP_007.pdf